CLINICAL TRIAL: NCT05463588
Title: The Effect of Exercise Conducted With Virtual Reality Glasses on Pain, Daily Life Activities and Quality of Life In Individuals With Lumbar Disc Herniation
Brief Title: Individuals With Lumbar Disc Hernia Exercising With Virtual Reality Glasses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, serap BUZTEPE, lead researcher, Ataturk University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: Atatürk university-001
Record Dates: First submitted 2022-07-08; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: To Evaluate the Effect of Exercise With Virtual Glasses on Pain, Activities of Daily Living and Quality of Life
Keywords: lumbar disc herniation; virtual reality glasses; pain; quality of life; activities of daily living
MeSH Terms: conditions — Intervertebral Disc Displacement; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Collection of pre-test data from the experimental and control groups (Experimental): Asking vas, ODI, sf-36 quality of life scale questions
  Interventions: Other: Exercising with virtual reality glasses
- Calculation of the pre-test fall risk index (Experimental): Calculation of patients' fall risk indices
  Interventions: Other: Exercising with virtual reality glasses
- giving back health education to the experimental and control groups (Experimental): Back health training was given to both groups, and the experimental group was given training on using virtual glasses.
  Interventions: Other: Exercising with virtual reality glasses
- collection of post-test data for the experimental and control group (Experimental): Asking vas, ODI, sf-36 quality of life scale questions
  Interventions: Other: Exercising with virtual reality glasses
- Calculation of the post-test fall risk index (Experimental): Calculation of patients' fall risk indices
  Interventions: Other: Exercising with virtual reality glasses

INTERVENTIONS:
Other: Exercising with virtual reality glasses — GIVE PATIENTS EXERCISE WITH A 360 DEGREE EXERCISE VIDEO INSIDE VIRTUAL REALITY EYES.
  Exercising with the training material taught at the beginning of the training
  Other Names: Exercising without virtual reality glasses

SUMMARY:
The purpose of this research; exercise performed with virtual reality glasses for individuals with lumbar disc herniation; The aim of this study is to examine the effects on pain, activities of daily living, quality of life and falling.

DETAILED DESCRIPTION:
The purpose of this research; exercise performed with virtual reality glasses for individuals with lumbar disc herniation; The aim of this study is to examine the effects on pain, activities of daily living, quality of life and falling.

This research was carried out experimentally with pretest-posttest control group.

The research was carried out between December 2019 and August 2022. The research was carried out in the Physical Therapy Unit of Erzurum Atatürk University Health Practice and Research Center.

The universe of the research; It consisted of 68 patients with LDH who came to Atatürk University Health Application and Research Center Physical Therapy and Rehabilitation Unit between 13 September 2022 and 7 January 2022.

n data collection, "Patient Identification Form" (Appendix-5), "Visual Analog Scale" (Appendix-6), "Oswestry Disability Index" (Appendix-7), "SF-36 Quality of Life Scale" (Appendix-8) and Falling Risk Score result is used.The patients in the experimental and control groups were first given training on protection of back health and exercise.

The patients in the experimental group did waist exercises with virtual reality glasses for 2 sessions, 28 sessions in total, every weekday.

ELIGIBILITY:
Inclusion Criteria:

* Being literate.
* Not having a physical disability that prevents them from doing the exercises.
* Not have an uncontrolled chronic or acute illness.
* Not having a vision problem that cannot be controlled by assistive methods.
* Not having a vertigo problem
* To be cognitively competent.
* Not having any musculoskeletal surgery in the last 6 months
* Not having knee joint disease
* To be able to complete the measurement with the balance device
* Having a body mass index below 40

Exclusion Criteria:

* To have a medium and high fall risk score in the measurement made with the balance device
* Experiencing chronic pain.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
Filling in the Visual Analog scale form before the intervention fort the LDH patients icluded in the study | Before starting the first treatment in the physical therapy unit (first day)
  The minimum score to be taken is 0 and the maximum score is 10. İt is known that as the score obtained increases,the pain felt by the patient increases
Filling in the SF-36 Ouality of life scale form before the intervention fort the LDH patients icluded in the study | Before starting the first treatment in the physical therapy unit (first day)
  The minimum score obtained from the SF-36 quality of life scale is 0 and the maximum score is 100. The higher the score, the higher the patient's quality of life
Filling in the Oswestry Disability Index form before the intervention fort the LDH patients icluded in the study | Before starting the first treatment in the physical therapy unit (first day)
  The minimum score obtained from the Oswestry Disability Index is 0 and the maximum score is 50. The lower the score, the greater the independence of the patient in his daily activities
Calculation of the fall risk index based on % points before the intervention fort he LDH patients included in the study | Before starting the first treatment in the physical therapy unit (first day)
  The lowest score to be taken from the risk index is 0 and the highest score is 100. The lower the Score received, the lower the risk

SECONDARY OUTCOMES:
Filling the Visual Analog scale form for LDH patients who have completed their 3-week intervention | After 3 weeks of intervention
  The minimum score to be taken is 0 and the maximum score is 10. İt is known that as the score obtained increases,the pain felt by the patient increases
Filling the Oswestry Disability Index form for LDH patients who have completed their 3-week intervention | After 3 weeks of intervention
  The minimum score obtained from the Oswestry Disability Index is 0 and the maximum score is 50. The lower the score, the greater the independence of the patient in his daily activities
Filling the SF-36 Ouality of life scale form for LDH patients who have completed their 3-week intervention | After 3 weeks of intervention
  The minimum score obtained from the SF-36 quality of life scale is 0 and the maximum score is 100. The higher the score, the higher the patient's quality of life
Calculation of the fall risk index of LDH patients over % points after 3 weeks of intervention | After 3 weeks of intervention
  The lowest score to be taken from the risk index is 0 and the highest score is 100. The lower the Score received, the lower the risk

CONTACTS AND LOCATIONS:
Locations (1):
- serap Buztepe, Erzurum, Palandöken, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buztepe S, Capik C. The effect of exercises done with virtual reality glasses on pain, daily life activities, and quality of life of individuals with lumbar disc hernia: a randomized controlled trial. BMC Musculoskelet Disord. 2025 Oct 1;26(1):886. doi: 10.1186/s12891-025-09130-9. PMID 41029303